CLINICAL TRIAL: NCT00992641
Title: The Effect of Nordic Diet Rich in Whole Grain, Berries, Fruits, Vegetables and Fish on Features of Metabolic Syndrome - a Systems Biology Approach
Brief Title: The Effect of Nordic Recommended Diet on the Features of Metabolic Syndrome - Multicentre Study
Acronym: SYSDIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: University of Copenhagen (Other); Aarhus University Hospital (Other); University of Oulu (Other); University of Iceland (Other); Oslo and Akershus University College (Other); Uppsala University (Other); Lund University (Other)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSDIET 070014; 31//2009
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Abdominal Obesity; Insulin Resistance; Impaired Glucose Tolerance; Type 2 Diabetes; Cardiovascular Diseases
Keywords: Systems biology; Nutrition; Nordic diet; Dietary recommendations; Metabolic syndrome; Features of metabolic syndrome
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance; Glucose Intolerance; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental diet (Experimental): Diet based on Nordic recommendations: rich in whole grain products, berries, fruits and vegetables, recommended fat quality. Realised based on eating habits of each Nordic country.
  Interventions: Other: Experimental diet
- Control diet (Active Comparator): Diet based on the information of the current dietary intake and food consumption in Nordic countries.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Experimental diet — Diet based on Nordic recommendations: rich in whole grain products, berries, fruits and vegetables, recommended fat quality. Realised based on eating habits of each Nordic country.
  Arms: Experimental diet
Other: Control diet — Diet based on the information of the current dietary intake and food consumption in Nordic countries.
  Arms: Control diet

SUMMARY:
SYSDIET (Systems biology in controlled dietary interventions and cohort studies) is one of the three centres in the NCoE Food, Nutrition and Health, 2007-2011. It consists of 12 partners from five Nordic countries working on multidisciplinary fields of science related to nutritional biology. The main objective of SYSDIET is to reveal mechanisms by which Nordic foods and diets could be modified to promote health and prevent insulin resistance, type 2 diabetes and cardiovascular diseases, all of which being connected to metabolic syndrome. Furthermore, the aim is to build up a Nordic platform for cohort studies and carefully conducted multi-centre dietary intervention studies, where novel nutritional systems biology tools can be applied besides human studies also in animal and cell culture studies. In order to achieve the main objective a Nordic multi-centre randomized controlled human intervention study is being conducted in 2009-2010 in 6-8 centres of SYSDIET consortium.

Health of the Nordic populations has substantially improved during the last 30 years. This is due e.g. to marked decline in cardiovascular morbidity and mortality. However, during the last 10-20 years increasing obesity and sedentary lifestyle have resulted in an increase of metabolic syndrome and type 2 diabetes.

Having this background, the aim of the SYSDIET consortium is to carry out a controlled, randomized dietary intervention study in persons with features of metabolic syndrome to find out the effects of a healthy Nordic food on major abnormalities in metabolic syndrome.

Altogether 167 persons aged 30 to 65 years were recruited from 6-8 centers (40-60 subjects/center) of the SYSDIET cohort. The main inclusion criterion is BMI 27-38 kg/m2. The subjects should also have at least two other IDF criteria for metabolic syndrome. Recruited persons will start the study by following their conventional diet for one month as a run-in period. After that subjects will be randomly assigned into Experimental- or Control-diet-group for 6 months. Experimental diet is rich in whole grain products, berries, fruits, vegetables and fish, and its fat intake is modified according to current Nordic recommendations. Control diet is based on the current information of the mean dietary intake and food consumption. The diets will be realized according to eating habits in each Nordic country.

DETAILED DESCRIPTION:
Substudy of the multicentre SYSDIET-study has been conducted in one of the centres, Aarhus, Denmark.

This study aims was determine if a "Healthy Nordic Diet (HND)" fulfilling the Nordic Nutrition Recommendations does affect 24-h ambulatory BP in subjects with features of Metabolic Syndrome. Of the 167 SYSDIET subjects with MeS, 37 were enrolled in a Danish sub study on 24-h ambulatory BP performed at 0 and 12 wks after randomization. 32 completed the sub study. All maintained stable body weight, physical activity level, medicine, and alcohol habits during the intervention, as prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 years old
* BMI 27-38 kg/m2
* + two other IDF criteria for metabolic syndrome
* Anti-hypertensives and lipid-lowering medication are allowed

Exclusion Criteria:

* Fasting plasma glucose > 7.0 mmol/l
* Fasting plasma triglycerides > 3.0 mmol/l
* Fasting plasma total cholesterol > 6.5 mmol/l
* Blood pressure > 160/100 mmHg
* Preceding weight change of 5% or more or active weight loss during preceding 6 months
* Any disease or condition that may hamper the successful participation of the intervention: liver disease, kidney disease, diabetes (both type 1 and type 2), thyroid disease (Newly found unstabilized disease), Myocardial infarction within previous 6 months
* Alcohol abuse (> 40 g/day)
* Oral corticosteroid therapy
* Severe psychiatric disorders
* Cancer under treatment
* Coeliac disease
* Exceptional diets (Atkin's, vegan, allergies to fish or cereals, other extensive allergies)
* Binge eating
* Unwillingness to discontinue the use of fish and vegetable oil or stanol and sterol ester supplements or products

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism | Study weeks 0
Glucose metabolism | 12 weeks
Glucose metabolism | 24 weeks

SECONDARY OUTCOMES:
Transcriptomics and metabolomics data | Study week 0
Transcriptomics and metabolomics data | 12 weeks
Transcriptomics and metabolomics data | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Dragsted, Prof, Principal Investigator — University of Copenhagen; Kjeld Hermansen, Prof, Principal Investigator — Aarhus University Hospital, Denmark; Kaisa Poutanen, Prof, Study Director — University of Kuopio, Finland; Matti Uusitupa, Prof, Study Director — University of Kuopio, Finland; Inga Thorsdottir, Prof, Principal Investigator — University of Iceland, Iceland; Markku Savolainen, Prof, Principal Investigator — University of Oulu, Finland; Karl-Heinz Herzig, Prof, Principal Investigator — University of Oulu, Finland; Stine M Ulven, Assoc prof, Principal Investigator — Akershus University College, Norway; Ulf Riserus, Prof, Principal Investigator — Uppsala University, Sweden; Björn Åkesson, Prof, Principal Investigator — Lund University; Peter Arner, Prof, Principal Investigator — Karolinska Institutet; Matej Oresic, Prof, Principal Investigator — VTT Technical Research Centre, Finland; Kim Overvad, Prof, Principal Investigator — Aalborg Hospital, Denmark; Carsten Carlberg, Prof, Principal Investigator — University of Kuopio, Finland; Grether I Borge, Senior Scientist, Principal Investigator — Nofima Foods, Norway
Locations (8):
- Denmark (2):
  - Aarhus University, Aarhus
  - University of Copenhagen, Copenhagen
- Finland (2):
  - University of Kuopio, Kuopio
  - University of Oulu, Oulu
- University of Iceland, Reykjavik, Iceland
- Akershus University College, Akershus, Norway
- Sweden (2):
  - Lund University, Lund
  - Uppsala University, Uppsala

REFERENCES:
- [Derived] Gurdeniz G, Uusitupa M, Hermansen K, Savolainen MJ, Schwab U, Kolehmainen M, Brader L, Cloetens L, Herzig KH, Hukkanen J, Rosqvist F, Ulven SM, Gunnarsdottir I, Thorsdottir I, Oresic M, Poutanen KS, Riserus U, Akesson B, Dragsted LO. Analysis of the SYSDIET Healthy Nordic Diet randomized trial based on metabolic profiling reveal beneficial effects on glucose metabolism and blood lipids. Clin Nutr. 2022 Feb;41(2):441-451. doi: 10.1016/j.clnu.2021.12.031. Epub 2021 Dec 25. PMID 35007813
- [Derived] Tuomainen M, Karkkainen O, Leppanen J, Auriola S, Lehtonen M, Savolainen MJ, Hermansen K, Riserus U, Akesson B, Thorsdottir I, Kolehmainen M, Uusitupa M, Poutanen K, Schwab U, Hanhineva K. Quantitative assessment of betainized compounds and associations with dietary and metabolic biomarkers in the randomized study of the healthy Nordic diet (SYSDIET). Am J Clin Nutr. 2019 Nov 1;110(5):1108-1118. doi: 10.1093/ajcn/nqz179. PMID 31504116
- [Derived] Lankinen M, Schwab U, Kolehmainen M, Paananen J, Nygren H, Seppanen-Laakso T, Poutanen K, Hyotylainen T, Riserus U, Savolainen MJ, Hukkanen J, Brader L, Marklund M, Rosqvist F, Hermansen K, Cloetens L, Onning G, Thorsdottir I, Gunnarsdottir I, Akesson B, Dragsted LO, Uusitupa M, Oresic M. A Healthy Nordic Diet Alters the Plasma Lipidomic Profile in Adults with Features of Metabolic Syndrome in a Multicenter Randomized Dietary Intervention. J Nutr. 2015 Apr 1;146(4):662-672. doi: 10.3945/jn.115.220459. PMID 26962194
- [Derived] Kolehmainen M, Ulven SM, Paananen J, de Mello V, Schwab U, Carlberg C, Myhrstad M, Pihlajamaki J, Dungner E, Sjolin E, Gunnarsdottir I, Cloetens L, Landin-Olsson M, Akesson B, Rosqvist F, Hukkanen J, Herzig KH, Dragsted LO, Savolainen MJ, Brader L, Hermansen K, Riserus U, Thorsdottir I, Poutanen KS, Uusitupa M, Arner P, Dahlman I. Healthy Nordic diet downregulates the expression of genes involved in inflammation in subcutaneous adipose tissue in individuals with features of the metabolic syndrome. Am J Clin Nutr. 2015 Jan;101(1):228-39. doi: 10.3945/ajcn.114.092783. Epub 2014 Nov 19. PMID 25527767
- [Derived] Magnusdottir OK, Landberg R, Gunnarsdottir I, Cloetens L, Akesson B, Rosqvist F, Schwab U, Herzig KH, Hukkanen J, Savolainen MJ, Brader L, Hermansen K, Kolehmainen M, Poutanen K, Uusitupa M, Riserus U, Thorsdottir I. Whole grain rye intake, reflected by a biomarker, is associated with favorable blood lipid outcomes in subjects with the metabolic syndrome--a randomized study. PLoS One. 2014 Oct 23;9(10):e110827. doi: 10.1371/journal.pone.0110827. eCollection 2014. PMID 25340768
- [Derived] Marklund M, Magnusdottir OK, Rosqvist F, Cloetens L, Landberg R, Kolehmainen M, Brader L, Hermansen K, Poutanen KS, Herzig KH, Hukkanen J, Savolainen MJ, Dragsted LO, Schwab U, Paananen J, Uusitupa M, Akesson B, Thorsdottir I, Riserus U. A dietary biomarker approach captures compliance and cardiometabolic effects of a healthy Nordic diet in individuals with metabolic syndrome. J Nutr. 2014 Oct;144(10):1642-9. doi: 10.3945/jn.114.193771. Epub 2014 Jul 30. PMID 25080537
- [Derived] Uusitupa M, Hermansen K, Savolainen MJ, Schwab U, Kolehmainen M, Brader L, Mortensen LS, Cloetens L, Johansson-Persson A, Onning G, Landin-Olsson M, Herzig KH, Hukkanen J, Rosqvist F, Iggman D, Paananen J, Pulkki KJ, Siloaho M, Dragsted L, Barri T, Overvad K, Bach Knudsen KE, Hedemann MS, Arner P, Dahlman I, Borge GI, Baardseth P, Ulven SM, Gunnarsdottir I, Jonsdottir S, Thorsdottir I, Oresic M, Poutanen KS, Riserus U, Akesson B. Effects of an isocaloric healthy Nordic diet on insulin sensitivity, lipid profile and inflammation markers in metabolic syndrome -- a randomized study (SYSDIET). J Intern Med. 2013 Jul;274(1):52-66. doi: 10.1111/joim.12044. Epub 2013 Mar 2. PMID 23398528
- See also: NCoE SYSDIET internet pages — http://www.sysdiet.fi/